CLINICAL TRIAL: NCT02189044
Title: Effects of the Method Pilates Exercises in Muscle Strength Respiratory of Elderly Women: a Clinical Trial
Brief Title: Pilates and Muscle Strength Respiratory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Lislei Jorge Patrizzi, Phd, Universidade Federal do Triangulo Mineiro
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UFTM2014
Record Dates: First submitted 2014-06-15; First posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Conditions
Keywords: aged;; breathing exercises;; muscle strength.
MeSH Terms: conditions — Disease | interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercises; muscle strength (Other): Evaluate the effects of Pilates exercises on respiratory muscle strength in elderly women before and after eleven weeks of training
  Interventions: Other: Pilates Exercise

INTERVENTIONS:
Other: Pilates Exercise — The training through the Pilates exercises were performed in eleven weeks. Each class consisted of five exercises lasting 40 minutes each lesson.
  During the first four weeks exercises performed were: Cat, Coffee Table, Single legcircle, pelvic movements, contraction of the glutes and closure was performed with posterior chain elongation range.
  In the next four weeks began a new series of exercises, which are: Bridge, Side Table, Bridge hip roll with legextension, Abdominal - halfhollup, obliques, and ultimately Stretching - Series of William's.
  In the last four weeks of training proposed a new series of exercises involving: Beaststroke, Support heel Bridge - hip roll with leg extension, and Hundred Squats with bat on the wall.

SUMMARY:
Introduction: Among the systems of the organism, it is believed that the respiratory system is the one which gets older faster due to the greater exposure to environmental pollutants over the years.The Pilates method has emerged as a form of fitness particularly providing general welfare to the individual. Objective: To evaluate the effects of Pilates' exercises on respiratory muscle strength in elderly women. Methods: The investigators have studied 07 women aged 60 and over, with preserved autonomy and cognitive skills. The Pulmonary Function Test (Spirometry) was performed using the Vitalograph® spirometer, model 8600. Respiratory muscle strength was obtained by technical measurements of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), through an analog Gerar manometer. The experiment lasted eleven (11) weeks. For comparative analysis of the data obtained in the evaluations, the investigators applied the paired t test and a significance level of 5%.

DETAILED DESCRIPTION:
METHODOLOGY This study is a clinical, longitudinal, prospective trial conducted at the Laboratory of Kinesiology and Cinesioterapia of Physiotherapy, Federal University of Triangulo Mineiro - UFTM. All participants signed an informed consent. The research started after approval by the Ethics Committee UFTM Research Protocol (2147-2012).

Subject Initially the invitation was made to all students enrolled in the Open University of Third Age - UATI / UFTM from August to October 2012.

The selection was based on the following inclusion criteria: (1) age and above 60 years, (2) non-practicing regular physical activity, (3) availability to attend Pilates classes twice a week (in addition to the time UATI ) and (4) with preserved cognitive autonomy and exclusion criteria: history (1) diseases that directly affect the posture (disc herniation and angular deformities of the spine), (2) cardiovascular, respiratory and neurological diseases that prevent attainment of Pilates exercises, (3) impaired cognitive capacity limited autonomy or self-determination, (4) withdrawal of participation during the assessment process, and (5) two consecutive absences or a total of three absences during the proposed time for the training set.

Thus, the proposed methodology for this study was applied in seven women with a mean age of 64 ± 6 years.

Review / Procedures The assessment instruments were used: (1) Initial Assessment Sheet, (2) spirometer and (3) manometer.

The record initial assessment and spirometry were applied for the selection of participants. Through the initial evaluation form was possible to assess aspects of health status of participants (associated diseases, blood pressure, respiratory and heart rate, postural assessment) as well as information on personal history, family history and current medication .

A pulmonary function test (spirometry) was performed using the Vitalograph ® spirometer brand model 8600. Equipment was calibrated, and the tests were performed by a single trained and qualified examiner with instructions and standardized voice commands, as I standards advocated by Consensus Brazilian on Espirometria.12 Spirometry was performed to rule out any lung disease that affects the performance of the proposed exercises.

To assess respiratory muscle strength, the volunteers remained in the standing position using a nose clip. Respiratory muscle strength was obtained by the techniques of measurements of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP), by means of an analog manometer Generate brand, scaled to ± 300 cmH2O, equipped with nozzle adapter, containing a hole 2 mm in diameter, serving as relief of muscles bocais.4 MIP valve was obtained with the maximal inspiration preceded by maximal expiration to residual volume level and MEP through the maximal expiration preceded by a maximal inspiration, to total lung capacity. Were performed at least three maneuvers maximal inspiratory pressure and maximal expiratory pressure, in order to obtain the greatest value from three acceptable.

The measurement of respiratory muscle strength occurred through an analog manometer (Ger-Air ®, São Paulo, Brazil), with scales - 300 to +300 cmH2O (calibrated), equipped with plastic trachea 16 cm long and 2.4 cm internal diameter, hard plastic mouthpiece and drain hole approximately 2 mm in diameter to dissipate the pressures generated by the muscles of the face and orofaringe.13 the maximal inspiratory pressure (MIP) and expiratory pressures were obtained maximum (MEP), carried a maximum of five times, acceptable and reproducible, and in the standing position, using a nose clip, for a time of sustained three seconds. The value of MIP was obtained from residual volume, and MEP from total lung capacity. Volunteers were due verbal encouragement and if there were more than 10% between a measure and another, a new difference maneuver was performed, considering the highest value since this was not the último.14 Therapeutic Intervention - Pilates Method The training through the Pilates exercises were performed in eleven weeks. The participants were instructed not to miss and attend classes twice a week. Each class consisted of five exercises lasting 40 minutes each lesson.

During the first four weeks (1 st to 4 th week) exercises performed were: Cat, Coffee Table, Single legcircle, pelvic movements, contraction of the glutes and closure was performed with posterior chain elongation range.

In the next four weeks (5th to 8th weeks) began a new series of exercises, which are: Bridge, Side Table, Bridge hip roll with legextension, Abdominal - halfhollup, obliques, and ultimately Stretching - Series of William's.

In the last four weeks of training (9th to 11th weeks) proposed a new series of exercises involving: Beaststroke, Support heel Bridge - hip roll with leg extension, and Hundred Squats with bat on the wall.

All exercises were performed during expiration. Statistical Analysis Descriptive data analysis was performed, with a mean and standard deviation. For comparative analysis of the data obtained in the pre-and post-intervention, the paired t test was applied (after confirmed the normal distribution of the sample - Shapiro Wilk test). The level of significance was set at 5%. The statistical program used was 18.0 SSPSS.

ELIGIBILITY:
Inclusion Criteria:

* age and above 60 years,
* non-practicing regular physical activity
* availability to attend Pilates classes twice a week (in addition to the time UATI)
* with preserved cognitive autonomy

Exclusion Criteria:

* history of diseases that directly affect the posture (disc herniation and angular deformities of the spine)
* cardiovascular, respiratory and neurological diseases that prevent attainment of Pilates exercises
* impaired cognitive autonomy or limited capacity for self-determination
* withdrawal of participation during the assessment process
* two consecutive absences or a total of three absences during the proposed training set for the time.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test (spirometry). | The results were obtained at the end of the eleven weeks of intervention

SECONDARY OUTCOMES:
Respiratory muscle strength | The results were obtained at the end of the eleven weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lislei Patrizzi, Principal Investigator — Universidade Federal do Triângulo Mineiro
Locations (1):
- Lislei Jorge Patrizzi, Uberaba, Minas Gerais, Brazil